CLINICAL TRIAL: NCT05747118
Title: A Feasibility Study of a 12 Week Training Intervention With Patients With Type 2 Diabetes and MODY in Greenland
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Greenland (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Maja Hykkelbjerg Nielsen, MSc in Public Health, PhD student, Steno Diabetes Center Greenland
Other Study IDs: 2022-21
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; MODY
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Physical Conditioning, Human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: People with type 2 diabetes or MODY in the training group
  Interventions: Behavioral: Physical training
- Control: People with type 2 diabetes or MODY in the control group

INTERVENTIONS:
Behavioral: Physical training — A 12 week supervised training intervention with 1 hour physical training two times a week.
  Groups: Intervention

SUMMARY:
The goal of this study is to investigate to what extent a 12-week training course for people with type 2 diabetes mellitus (T2DM) or MODY can be conducted in a clinical context with clinically relevant improvements in cardiometabolic risk factors and quality of life?

The main questions it aims to answer are:

1. To investigate the feasibility of supervised training for people with T2DM or MODY in a clinical context in Greenland.
2. To investigate evidence of the effect of combined aerobic and strength training on cardiometabolic risk factors and mental well-being.
3. To investigate the signs of efficacy and different interactions with the type of disease.

DETAILED DESCRIPTION:
Globally, type 2 diabetes mellitus (T2DM) is a major public health issue. This is also the fact in Greenland, the biggest island in the world.

Twice as many Greenlanders as Danes have diabetes, and this is due to both lifestyle and genes. It is estimated that 7% of T2DM patients in Greenland have Maturity Onset Diabetes of the Young (MODY), which is hereditary and rare elsewhere.

Exercise improves blood sugar control in T2DM, reduces cardiovascular risk factors such as hypertension and dyslipidemia, contributes to weight loss and improves fitness and well-being. Less is known of how people with MODY responds to exercise.

Today, the Greenlandic health care system only offers supervised physical training to people with osteoarthritis in two towns in Greenland, but in the future, they would like to offer supervised physical training to people with other conditions too.

Relevance: As mentioned above, this study aims to evaluate the feasibility of a 12-week supervised physical training intervention for people with T2DM or MODY and to investigate signs of efficacy and different interactions with the type of disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes or MODY
* Living in the capital in Greenland, Nuuk

Exclusion Criteria:

* Severe heart disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants were recruited within the Capital of Greenland, Nuuk. Males and females >18 years old and diagnosed with T2DM or MODY were included. The exclusion criteria were severe heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence | Baseline to 12 weeks
  Adherence is in this study the proportion of completed training sessions (n=0-24 training sessions). The number of completed training sessions was registered by the physiotherapists.

SECONDARY OUTCOMES:
Change in quality of life | Baseline to 12 weeks
  Quality of life is estimated using 12-Item Short Form Survey (SF-12). In the short form SF-12, physical (SF12-PCS) and mental (SF12-MCS) component summary scores are calculated as sub-dimensions. The total score of the physical and mental component summary of the scale varies between 0-100. An increase in the score indicates well-being, and a decrease indicates a state of disability.
Change in BMI | Baseline to 12 weeks
  BMI is measured using height and weight.
Change in fat mass | Baseline to 12 weeks
  Fat mass is measured using tanita body composition analyzer.
Change in muscle mass | Baseline to 12 weeks
  Muscle mass is measured using tanita body composition analyzer.
Change in bone mass | Baseline to 12 weeks
  Bone mass is measured using tanita body composition analyzer.
Change in blood pressure | Baseline to 12 weeks
  Blood pressure is measured with a blood pressure monitor.
Change in HbA1c | Baseline to 12 weeks
  HbA1c is measured with a blood sample.
Change in HDL cholesterol | Baseline to 12 weeks
  HDL cholesterol is measured with a blood sample.
Change in LDL cholesterol | Baseline to 12 weeks
  LDL cholesterol is measured with a blood sample.
Change in Total cholesterol | Baseline to 12 weeks
  Total cholesterol is measured with a blood sample.
Change in triglycerides | Baseline to 12 weeks
  Triglycerides is measured with a blood sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Greenland, Nuuk, Greenland

IPD SHARING:
Plan to Share IPD: No